CLINICAL TRIAL: NCT00372294
Title: To Compare Intravitreal Clindamycin & Dexamethasone With Classic Treatment of Toxoplasmic Retinochoroiditis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8415
Record Dates: First submitted 2006-09-05; First posted 2006-09-06 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2008-06

CONDITIONS: Chorioretinitis
Keywords: Toxoplasmosis; Chorioretinitis; Intravitreal Clindamycin; Dexamethasone in chorioretinitis; Toxoplasmic
MeSH Terms: conditions — Chorioretinitis; Toxoplasmosis | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Active Comparator): Classic regimen (Pyrimethamine-Sulfadiazine + Prednisolon)
  Interventions: Drug: pyrimethamine-sulfadiazine + prednisolone
- 2 (Active Comparator): Intravitreal Clindamycin & Dexamethasone
  Interventions: Drug: Clindamycin+Dexamethasone

INTERVENTIONS:
Drug: pyrimethamine-sulfadiazine + prednisolone — Administration of pyrimethamine-sulfadiazine + prednisolone
  Arms: 1
Drug: Clindamycin+Dexamethasone — Intravitreal injection of Clindamycin+Dexamethasone
  Arms: 2

SUMMARY:
Toxoplasmosis, an intra cellular parasite, is a very important cause of chorioretinitis. The goal of treatment is arresting multiplication of the parasite in its inflammatory active phase. In this study the investigators try to compare the efficacy of the classic regimen (Pyrimethamine-Sulfadiazine + Prednisolon) with intravitreal Clindamycin & Dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Toxoplasmic chorioretinitis
* Location of the lesion within zone I of the retina or a lesion greater than 2DD with 3+-4+ vitreous inflammation in zone II or III
* No allergic history to the used drugs
* No any other diseases

Exclusion Criteria:

* Any allergic reaction to the used medications
* One eyed patients
* Partially treated patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-07; Primary Completion 2008-08 (Estimated); Study Completion 2008-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Masoud Soheilian, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Ophthalmic Research Center, Tehran, Tehran Province, Iran